CLINICAL TRIAL: NCT05203783
Title: Short-term Effects of Kinesio Taping in Patients With Mechanical Low Back Pain: A Randomized Clinical Trial.
Brief Title: Short-term Effects of Kinesio Taping in Patients With Mechanical Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Eren Timurtas, Principal Investigator, Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-1039
Record Dates: First submitted 2022-01-21; First posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): The control group will receive only McKenzie exercises for 7 days.
  Interventions: Other: McKenzie Exercises; Other: Kinesio Tape Application
- Experimental Group (Experimental): The experimental group will receive Kinesio tape application in addition to McKenzie exercises for 7 days.
  Interventions: Other: Kinesio Tape Application

INTERVENTIONS:
Other: McKenzie Exercises — McKenzie exercises: The McKenzie set consists of 5 exercises.
  1. Prone-lying
  2. Prone-extension
  3. Prone press ups
  4. Progressive extension with pillows
  5. Standing extension
  Arms: Control Group
Other: Kinesio Tape Application — Kinesio Tape (KT) application: Participants in the experimental group received additional taping using KT by an experience therapist with prior training in KT application. The tape was applied using the method proposed for the sacrospinalis muscle (Kase, 1996). Y-shaped tape was applied as shown in Figure 1. While the participant was in standing position, the origin of the Y-shaped tape was attached over the centre of the sacrum without stretching the tape and afterward subjects gradually bent forward. A 5-degree angle was maintained within the valley of the Y tape. The tape was changed on the fourth day

SUMMARY:
The aim of this study is to estimate the effect of Kinesio tape (KT) combined with supervised exercise programs compared to exercise alone on pain, lumbar range of motion, and self-reported disability of adults with mechanical low back pain (LBP).

Methods: This was a randomized, controlled clinical trial carried out on 60 individuals with mechanical LBP. Participants were randomly assigned to the control group (n=30) that received McKenzie exercises for 7 days or experimental group (n=30) that received KT application in addition to McKenzie exercises for 7 days. Pain measured by visual analogue scale, lumbar range of motion, and the disability measured by Oswestry Disability Index (ODI) were used as outcome measures. Pre and Post measurements were taken at baseline and after 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with mechanical LBP by a physician

Exclusion Criteria:

* Individuals with any structural or pathological changes (spondylitis, spondylolisthesis, cauda equina syndrome, lumbar canal stenosis) in lumbar spine on X-ray or MRI
* Individuals with or without neurological signs in the lower extremity suggestive upper motor or lower motor neuron involvement,
* Individuals with a history of trauma or any surgery in the region of back,
* Individuals with recent aggravation of symptoms,
* Individuals on a waiting list for spinal surgery or had a spinal surgery in the past 6 months

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-08-08 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-25 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) | The pain was measured at baseline
  Pain was measured using a 10 cm visual analogue scale (VAS). The participants placed a mark on the line that best represented their perception of pain at that instant. The VAS score was measured in cm from the left hand end of the line to the mark.
Visual analogue scale (VAS) | The pain was measured at the end of intervention (7th day).
  Pain was measured using a 10 cm visual analogue scale (VAS). The participants placed a mark on the line that best represented their perception of pain at that instant. The VAS score was measured in cm from the left hand end of the line to the mark.

SECONDARY OUTCOMES:
The Oswestry Disability Index (ODI) | The ODI was measured at study entry 2 minutes after the pain assesment.
  The ODI was used to assess the disability. The ODI is a valid and reliable tool that measures functional disability. The scale consists of 10 sections, each section the total possible score is ranging from 0 to 5. After that, the entire score is multiplied by two to get a percentage.
The Oswestry Disability Index (ODI) | The ODI was measured at the end of intervention (7th day) 2 minutes after the pain assesment.
  The ODI was used to assess the disability. The ODI is a valid and reliable tool that measures functional disability. The scale consists of 10 sections, each section the total possible score is ranging from 0 to 5. After that, the entire score is multiplied by two to get a percentage.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No